CLINICAL TRIAL: NCT03712111
Title: Comparison of Vasopressor Boluses for Management of Hypotension After Spinal Anesthesia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, Assistant professor of anesthesia and critical care, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N-71-2018
Record Dates: First submitted 2018-10-16; First posted 2018-10-19 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Cesarean Section Complications; Spinal Anesthetic Toxicity
MeSH Terms: interventions — Norepinephrine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Norepinephrine 6 mcg (Experimental): Mothers in this group will receive a bolus of Norepinephrine 6 mcg for management of hypotensive episode after spinal anesthesia using Bupivacaine hydrochloride under prophylactic Norepinephrine infusion
  Interventions: Drug: Norepinephrine 6 mcg; Drug: Bupivacaine Hydrochloride; Drug: Norepinephrine infusion
- Norepinephrine 10 mcg (Active Comparator): Mothers in this group will receive a bolus of Norepinephrine 10 mcg for management of hypotensive episode after spinal anesthesia using Bupivacaine hydrochloride under prophylactic Norepinephrine infusion
  Interventions: Drug: Norepinephrine 10 mcg; Drug: Bupivacaine Hydrochloride; Drug: Norepinephrine infusion

INTERVENTIONS:
Drug: Norepinephrine 6 mcg — An intravenous bolus of norepinephrine 6 mcg will be administered for management of maternal hypotension.
  Other Names: Levophed
  Arms: Norepinephrine 6 mcg
Drug: Norepinephrine 10 mcg — An intravenous bolus of norepinephrine 10 mcg will be administered for management of maternal hypotension.
  Other Names: Levophed
  Arms: Norepinephrine 10 mcg
Drug: Bupivacaine Hydrochloride — Subarachnoid block will be performed using Bupivacaine hydrochloride (2.2 mL) in addition to fentanyl 25 mcg
  Other Names: Marcaine
Drug: Norepinephrine infusion — Prophylactic norepinephrine infusion will be started after subarachnoid block
  Other Names: Levophed

SUMMARY:
In this study the investigators will compare the efficacy and side effects of two doses of norepinephrine bolus (6 mcg and 10 mcg) in management of maternal hypotensive episode after subarachnoid block during Cesarean delivery.

DETAILED DESCRIPTION:
Maternal hypotension after subarachnoid block is a frequent and deleterious complication during cesarean delivery. Although prophylaxis against hypotension using vasopressors had become a standard recommendation; the incidence of hypotension is still ∼ 20% . Thus; management of maternal hypotension using vasopressor boluses is usually needed .

The commonly used vasopressors during cesarean delivery are ephedrine, phenylephrine, and recently norepinephrine. The use of ephedrine is usually accompanied with maternal tachycardia and fetal acidosis. Phenylephrine had been the first line for prevention and management of maternal hypotension; however, its use might result in bradycardia and decreased maternal cardiac output .

Norepinephrine is an alpha adrenergic agonist with weak beta adrenergic agonistic activity; thus, it does not cause significant cardiac depression as phenylephrine does. Norepinephrine was introduced for use during cesarean delivery with promising results . Few previous studies investigated the efficacy of Norepinephrine infusion for prevention of maternal hypotension. A dose-response study had investigated the best dose of Norepinephrine for prevention of maternal hypotension. In the aforementioned dose-response study, a dose of 6 mcg was reported as the best dose for prophylaxis against maternal hypotension.

No studies had investigated the best bolus dose of norepinephrine for management of a maternal hypotensive episode. In this study the investigators will investigate the efficacy and side effects of two doses of norepinephrine bolus doses (6 mcg and 10 mcg) in management of maternal hypotensive episode after subarachnoid block during cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* scheduled for cesarean delivery

Exclusion Criteria:

* patients with severe cardiac dysfunction
* patients with low blood pressure
* patients with ante-partum bleeding

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Estimated)
Dates: Start 2018-11-21 (Actual); Primary Completion 2022-06-25 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Rate of successful management of maternal hypotension | 30 minutes after spinal anesthesia
  number of patients with successful management of maternal hypotensive episode (defined as return of systolic blood pressure to be ≥ 80% of the baseline reading in the next reading 2 minutes after administration of norepinephrine bolus)

SECONDARY OUTCOMES:
Rate of successful management of severe maternal hypotension | 30 minutes after spinal anesthesia
  number of patients with successful management of maternal severe hypotensive episode (defined as systolic blood pressure lower than 60% of the baseline reading in the next reading 2 minutes after administration of norepinephrine bolus)
incidence of reactive hypertension | 30 minutes after spinal anesthesia
  number of patients with reactive hypertension (defined as systolic blood pressure ≥120% from the baseline reading after administration of norepinephrine bolus)
systolic blood pressure | 90 minutes after spinal anesthesia
  systolic blood pressure measured in mmHg
heart rate | 90 minutes after spinal block
  number of heart beats per minute
Apgar score for evaluation of the activity of the fetus | 10 minutes
  the Apgar score of the fetus which range from 0 to 10. Th minimum value is 0 and the maximum value is 10. The worst value is 0 and the best value is 10
Umbilical blood acidity | 10 minutes after delivery
  the measure of acidity or alkalinity of any solution on a logarithmic scale on which 7 is neutral, lower values are more acid and higher values more alkaline.
The frequency of vomiting | 90 minutes after spinal anesthesia
  The number of patients with vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Hasanin, Professor, Principal Investigator — Assistant professor of anesthesia
Locations (1):
- Ahmed Mohamed Hasanin, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No